CLINICAL TRIAL: NCT02687243
Title: Assessing the Effects of an Interactive Virtual Reality Intervention in Reducing Preoperative Anxiety in Children Undergoing Elective Surgery: A Randomized Controlled Trial Study Protocol
Brief Title: StoryTelling Medicine Application Using a Virtual Reality Intervention
Acronym: STM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-1220
Record Dates: First submitted 2016-01-15; First posted 2016-02-22 (Estimated); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Anxiety
Keywords: pediatrics; anxiety; anesthesia; preoperative
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive Virtual Application (Experimental): Online application
  Interventions: Device: Interactive Virtual Application
- Standard of Care (No Intervention): No intervention and Hospital Standard of Care

INTERVENTIONS:
Device: Interactive Virtual Application — Online application via tablet
  Arms: Interactive Virtual Application

SUMMARY:
Preoperative anxiety (PA) affects up to 5 million children in North America each year and is associated with adverse medical, psychological, and behavioral effects. Children who are highly anxious often require more medications during surgical procedures and take longer to recover. While many attempts have been made to reduce PA in children, existing interventions are limited by their expense and time intensive nature. Thus, the current lack of effective and efficient methods of reducing anxiety in children before and after surgery has prompted us to develop and propose to test a new intervention. The investigators have developed a novel,interactive tablet based Virtual Reality program, StoryTelling Medicine (STM), to help reduce anxiety in children undergoing elective surgery, and its associated negative effects.

STM is an age appropriate, customizable program to prepare children for complex surgical procedures by guiding them through the hospital settings. The investigators will examine if STM is effective in reducing PA and its adverse effects in children undergoing surgery. If effective, STM has the potential to improve children's and families' surgical experiences, and reduce health problems in the hospital setting and beyond.

DETAILED DESCRIPTION:
Children with PA not only suffer physically and emotionally, but some of them will develop fear of physicians and healthcare providers. These children tend to avoid future medical care and can lead to increased suffering for the child and their family, as well as higher rates of morbidity and health care costs.

There is a paucity of research evaluating the effects of AudioVisual interventions in reducing perioperative anxiety in children undergoing surgery. To date, no one has examined the physiological effects of PA or interventions designed to reduce it.

In the past 2 years, the investigators have conducted 3 pilot studies that have examined the stability of perioperative anxiety in children (n=90) and parents, as well as the feasibility of our recruitment and testing protocol, and to pilot test the interactive tablet-based application. The investigators have established that PA can be reliably and validly measured in children and that the rate of participant recruitment, data collection, website adherence and follow-up protocols for the proposed study are feasible and acceptable. The investigators will now progress to conduct the randomized controlled trial (RCT).

This RCT will be the first to examine the effects of STM in reducing PA and perioperative outcomes in children undergoing elective surgery. Therefore, the investigators will include both behavioral (i.e., observer- and self-rated) and biological measures of stress (i.e., heart rate, salivary cortisol) to further our understanding of the impact of STM on PA.

Unlike existing interventions, the customizable STM program provides a simulated hospital environment that can not only educate, but also increase children's coping abilities to better prepare them for surgery. In addition to reducing children's PA, it can also play an important role in reducing parental anxiety by preparing parents with a knowledge tool to support their child throughout the surgical process.The investigators believe that STM is a promising tool to improve children's health and ease the familial and societal costs of PA in an easy and cost-effective way. Given that many children in other hospitals do not receive adequate preoperative preparation, STM has the potential to provide proper perioperative care for every child in need.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 8-13 who are scheduled to receive any outpatient surgery (i.e. tonsillectomy, herniorrhaphy)

Exclusion Criteria:

* Children with chronic illnesses (e.g., cancer), known neurodevelopmental disorders, or who are on psychotropic medications prior to randomization will be excluded

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 118 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Preoperative anxiety | Baseline, Day 1 and One Month
Change in Heart rate | Baseline and Day 1
Change in Salivary Cortisol | Baseline and Day 1
  Saliva cortisol test in ng/dL

SECONDARY OUTCOMES:
Anesthetic induction compliance | Day 1
Anesthetic Dosage for Sedation | Day 1
  Anesthetic agent and dosage used
Delirium | Day 1
  Nursing notes
Length of Stay | Day 1
  Hospital records
Analgesic Usage | Day 1
  Medication Chart
Post-Hospital Behaviour | One month
  Using Post-Hospital Behaviour Questionnaire (PHBQ)

CONTACTS AND LOCATIONS:
Overall Officials: Desigen Reddy, MD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chow CH, Van Lieshout RJ, Schmidt LA, Dobson KG, Buckley N. Systematic Review: Audiovisual Interventions for Reducing Preoperative Anxiety in Children Undergoing Elective Surgery. J Pediatr Psychol. 2016 Mar;41(2):182-203. doi: 10.1093/jpepsy/jsv094. Epub 2015 Oct 17. PMID 26476281